CLINICAL TRIAL: NCT07330258
Title: A Natural History Study of Treated Parkinson's Disease Patients Experiencing Motor Complications
Brief Title: A US Study That Observes How Parkinson's Disease Changes Over Time in Patients Who Still Have Movement Symptoms Despite Taking Parkinson's Medications
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23021
Record Dates: First submitted 2025-12-09; First posted 2026-01-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
Keywords: Natural history study; Parkinson's disease; PD Motor (Hauser) Diary; MDS-UPDRS; Electronic health/medical records; Administrative claims data; Biological samples; Digital health technology; Care partner
MeSH Terms: conditions — Parkinson Disease | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (serum, plasma), Skin biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parkinson's Disease Cohort: A single cohort of patients with Parkinson's disease experiencing motor complications while receiving standard-of-care oral therapies. The care partner of the patient may also participate in the study.
  Interventions: Other: Standard of Care
- Care Partners Cohort: The care partner of the patient may also participate in the study.

INTERVENTIONS:
Other: Standard of Care — Follow clinical practice/administration. No investigational products will be administered in this study. Patients will be treated in accordance with standard of care as determined by their clinician.
  Groups: Parkinson's Disease Cohort

SUMMARY:
This is an observational study in which data are collected and studied from Parkinson's disease patients who have movement symptoms despite taking standard Parkinson's medications. In observational studies, observations are made without any changes to the participant's healthcare or treatment plan. No investigational product will be administered in this study, as participants will be treated with the standard of care that medical experts currently consider most appropriate.

Parkinson's disease (PD) is a condition that affects the brain and causes problems with movement and other body functions. The symptoms of Parkinson's disease can worsen over time. People with Parkinson's disease may experience shaking (tremor), slow movements, stiff muscles, trouble walking, and problems with balance. They can also have other symptoms, such as difficulty thinking clearly, changes in mood, or difficulty sleeping. Parkinson's disease mostly affects older adults, but it can happen to younger people too. There is no cure, but treatments can help manage the symptoms and improve quality of life.

While doctors and researchers know that Parkinson's disease affects people in different ways and can worsen over time, there are still many things they don't fully understand-especially for people who experience movement symptoms despite taking their usual Parkinson's medicines. Earlier studies did not follow these patients long enough or collect all the important information needed. This study is being done to fill those gaps.

The main purpose of this study is to better understand how Parkinson's disease changes over time in patients who experience movement symptoms while taking standard oral Parkinson's medications, what challenges patients and their care partners face, and how their treatments are working in real life. To do this, researchers will collect data on:

* Sociodemographics (e.g. age, gender, race/ethnicity, insurance provider).
* Medical history and vital signs (e.g. comorbidities, family history of Parkinson's, height, weight, blood pressure).
* Medications and treatments (e.g. Parkinson's and non-Parkinson's medications and other treatments, rehabilitation therapy sessions, use of mobility assistance devices).
* Movement symptoms (e.g. tremor, slow movement, balance).
* Non-movement symptoms (e.g. cognition, mood, sleep, activities of daily living).
* Molecular data (e.g. genetics, α-synuclein).
* Burden of care (e.g. economic cost).

Data will come from questionnaires or rating scales conducted by the doctor with the patient during study visits, diaries and logs completed by the patient, medical records, health insurance claims records, blood samples and skin biopsies, a digital device that records movement/non-movement symptoms, and questionnaires completed by the care partner.

Data will be collected from December 2025 to December 2032. Each participant may be followed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria for Patient:

* Individual of any sex ≥45 to ≤75 years of age at informed consent (at least 30% ≤60 years of age).
* Diagnosis of clinically established Parkinson's disease (PD) as defined by the Movement Disorder Society (MDS) Clinical Diagnostic Criteria for PD ≥4 and <12 years from time of PD diagnosis at informed consent.
* Modified H&Y stage II-III in the practically defined OFF-medication state (≥12 hours from last dose of antiparkinsonian medications).
* Score of ≥30 on MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III in the OFF-medication state.
* Presence of motor fluctuations with ≥1 hour of absolute time in the OFF state per day as assessed by clinician/patient at screening.
* Receiving stable antiparkinsonian medication regimen for ≥4 weeks prior to screening with a levodopa daily dose ≥300 mg or a dosing frequency of ≥3 times per day.
* Responsiveness to levodopa as determined by change in the following measures from the practically defined OFF state to ON state after taking typical first-daily dose of PD-medications: i. any degree of improvement (≥0.5 point) in modified H&Y stage OR. ii. ≥30% improvement in MDS-UPDRS part III score.
* Montreal Cognitive Assessment (MoCA) score of ≥24.
* Agree to participate and provide signed informed consent.

Exclusion Criteria for Patient:

* Known history or presence of conditions that may provide an alternative to a PD diagnosis including but not limited to: multiple system atrophy, progressive supranuclear palsy, striatonigral degeneration, corticobasal syndrome/degeneration, vascular Parkinsonism, drug-induced Parkinsonism, essential tremor, diffuse Lewy body disease, Lewy body dementia, Huntington's disease, Wilson's disease, Fahr's disease, Alzheimer's disease, cerebrovascular disease, brain tumor, trauma, and infection.
* Known history or presence of significant vascular and/or cardiovascular disease limited to: stroke, transient ischemic attacks, poorly controlled hypertension, poorly controlled diabetes, unstable angina pectoris, or unstable myocardial infarction.
* Known history or presence of significant psychosis or impulse control disorder, or untreated or sub optimally treated depression.
* Known history or presence of human immunodeficiency virus, hepatitis B virus, hepatitis C virus, syphilis, or tuberculosis.
* Current or previously active malignant disease within the past 5 years, except definitively treated cutaneous squamous cell carcinoma, basal cell carcinoma, or in situ uterine cervical carcinoma.
* Currently pregnant, nursing, lactating, breastfeeding, or plan to be during study duration.
* Known history or current use of percutaneous levodopa/carbidopa intestinal gel, subcutaneous levodopa, or apomorphine pump.
* Prior history of brain surgery, including but not limited to: deep brain stimulation (DBS), pallidotomy, focused ultrasound thalamotomy, or other experimental neurosurgical procedure.
* Known history or current participation in cell or gene therapy procedures.
* Current participation in any interventional clinical trial.

Inclusion Criteria for Care Partner:

* ≥18 years of age at informed consent.
* Identified by the PD patient as their primary care partner.
* Agree to participate and the ability to provide signed informed consent independently, without the need for a legal representative.

Exclusion Criteria for Care Partner:

* Not applicable.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease experiencing motor complications while on antiparkinsonian medications
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2032-12-01 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive summary of motor outcomes among Parkinson's disease patients treated with oral antiparkinsonian medications who experience motor complications. | From baseline up to 5 years
  This outcome will be assessed using Parkinson's disease (PD) Motor (Hauser) Diary, Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts II-IV (each part has several items scored from 0-normal to 4-severe; with higher scores indicating greater impairment), modified Hoehn & Yahr (stages Parkinson's disease severity from 1 [unilateral involvement only] to 5 [wheelchair-bound or bedridden unless aided]), Universal Dyskinesia Rating Scale (UDysRS) (items scored from 0-none to 4-severe; higher scores indicate more severe dyskinesia), medical records, and digital health technology.
Descriptive summary of non-motor outcomes among Parkinson's disease patients treated with oral antiparkinsonian medications who experience motor complications. | From baseline up to 5 years
  This outcome will be assessed using Montreal Cognitive Assessment (MoCA, score 0-30, higher = better cognition), MDS-UPDRS I (4-point scale, higher = greater impairment), modified Schwab & England Activities of Daily Living (0-100%, higher = greater independence), MDS Non-Motor Rating Scale (MDS-NMS, 4-point scale, higher = more severe non-motor symptoms), Parkinson's Disease Questionnaire-39 (PDQ-39, 0-100 scale, higher = worse quality of life), Parkinson's Disease Health Index (PD-HI, higher = worse health status), Parkinson's Disease Sleep Scale 2 (PDSS-2, 4-point scale, higher = more severe sleep problems), Clinical Global Impressions Severity (CGI-S, 7-point scale, higher = greater severity of illness), Patient Global Impression Severity (PGI-S, 7-point scale, higher = greater severity), EuroQoL 5-Dimension 5-Level (EQ-5D-5L, 5 dimensions, 5 levels, plus visual analogue scale (VAS) 0-100 [100=best imaginable health]), medical records, and digital health technology.
Descriptive summary of Parkinson's medications and treatments received | From baseline up to 5 years
  This outcome will be assessed by the logs (Parkinson's medications, Parkinson's advanced therapies, rehabilitation therapies & mobility assistance devices) completed by the patient, medical records, and health insurance claims records.
Descriptive summary on the burden of care - psychological dimension | From baseline up to 5 years
  This outcome will be assessed using the Zarit Burden Interview (ZBI), a 22-item questionnaire scored 0-88 (higher scores indicate greater burden).
Descriptive summary on the burden of care - economic dimension | From baseline up to 5 years
  This outcome will be assessed using the Caregiver Indirect and Informal Care Cost Assessment Questionnaire (CIIQ), which includes 13 questions on work status, productivity, and informal care costs.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - The Parkinson's & Movement Disorder Institute, Fountain Valley, California
  - Keck School of Medicine, Los Angeles, California
  - Boston University, Boston, Massachusetts
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.